CLINICAL TRIAL: NCT00150813
Title: A Multicenter, Open-label, Follow-up Trial Evaluating the Long-term Safety of Levetiracetam Individualized Dose From 1000 to 3000 mg/Day (Oral Tablets of 500 mg b.i.d.), Used as Monotherapy in Subjects (≥ 16 Years) Suffering From Epilepsy and Coming From the N01061 or the N01093 Trials.
Brief Title: Monotherapy With Levetiracetam in Patients Suffering From Epilepsy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01127
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2018-10-01 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-10

CONDITIONS: Epilepsy, Tonic-clonic
Keywords: Monotherapy; Epilepsy; Keppra; Levetiracetam
MeSH Terms: conditions — Epilepsy, Tonic-Clonic; Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Levetiracetam (Experimental): Subjects received open-label Levetiracetam.
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — Pharmaceutical form: oral tablets Route of administration: Oral use
  Other Names: Keppra

SUMMARY:
An open-label follow-up trial assessing the long term safety of levetiracetam as per adverse events reporting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a confirmed diagnosis of epilepsy.
* Subjects having experienced in the past unprovoked partial seizures (IA, IB, IC with clear focal origin),or generalized tonic-clonic seizures (without clear focal origin), that are classifiable according to the International Classification of Epileptic Seizures
* Subjects having participated in the previous double-blind monotherapy trial (N01061 [NCT00150735] or N01093 [NCT00150787]).
* Male/female subjects (>= 16 years).

Exclusion Criteria:

- Need for an additional Antiepileptic Drug (AED).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2005-08-10 (Actual); Primary Completion 2007-05-29 (Actual); Study Completion 2007-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (21):
- Czechia (5):
  - Beroun
  - Brno
  - České Budějovice
  - Prague
  - Rychnov nad Kněžnou
- Hungary (4):
  - Budapest
  - Debrecen
  - Pécs
  - Szeged
- Poland (7):
  - Bialystok
  - Gdansk
  - Katowice
  - Lodz
  - Lublin
  - Szczecin
  - Warsaw
- Sweden (5):
  - Gothenburg
  - Helsingborg
  - Huddinge
  - Karlstad
  - Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in August 2005 and concluded in May 2007.
Pre-assignment Details: Participant Flow refers to the Intention-to-Treat (ITT) Set.
Period: Overall Study
Arm/Group | Levetiracetam
Started | 66
Completed | 48
Not Completed | 18
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 5
Not completed — Remission | 3
Not completed — Planned pregancy | 1
Not completed — Switch to commercially available LEV | 2

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Intention-to-Treat (ITT) population.
Arm/Group | Levetiracetam
Number analyzed (Participants) | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 56
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.39 (18.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage Participants With Treatment Emergent Adverse Events
Description: An Adverse Event (AE) is any untoward medical occurrence (eg, noxious or pathological changes) in a subject or clinical investigation subject compared with pre-existing conditions, that occurs during any period of a clinical trial. An AE is defined as being independent of assumption of any causality (eg, to study or concomitant medication, primary or concomitant disease, or study design).
Time Frame: From the Entry Visit until up to 2 weeks after the last drug intake, up to 93 weeks
Population: Safety Set
Measure: Number; unit: percentage of participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 66
percentage of participants | 27.3

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the Entry Visit until up to 2 weeks after the last drug intake, up to 93 weeks.
Arm/Group | Levetiracetam
Serious Adverse Events (participants affected / at risk) | 4/66
Other Adverse Events (participants affected / at risk) | 0/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levetiracetam (N=66)
Encephalopathy (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Completed suicide (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days